CLINICAL TRIAL: NCT02546635
Title: A Safety, Tolerability, and Pharmacokinetic Clinical Trial of AX-024.HCl to Evaluate A) Potential Food Effect and B) Multi-dosing in Healthy Male Subjects
Brief Title: Potential Food Effect And Repeated Dosing of AX-024.HCl In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Artax Biopharma Inc (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: AX-024.HCl-1.02
Record Dates: First submitted 2015-08-11; First posted 2015-09-11 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potential food effect (Experimental)
  Interventions: Drug: AX-024.HCl
- Multi-dosing (Experimental)
  Interventions: Drug: AX-024.HCl

INTERVENTIONS:
Drug: AX-024.HCl — AX-024.HCl will be administered as per the protocol defined frequency and dose level
  Arms: Potential food effect
Drug: AX-024.HCl — AX-024.HCl will be administered as per the protocol defined frequency and dose level
  Arms: Multi-dosing

SUMMARY:
Part A: Food effect (a single oral dose of 500 mg AX-024.HCl under fasted and fed states) Eight (8) healthy male volunteers will receive a single dose of 500 mg AX-024.HCl in the fasted state (10 h overnight fast), and will return 2 weeks later to receive the same dose of AX-024.HCl following a meal.

Part B: Multiple doses (a once daily dose of AX-024.HCl or Placebo for 10 days).

Part B is a double-blind, dose escalating, placebo controlled, randomised, multiple dose study to assess the tolerability, safety and pharmacokinetics in 24 healthy male subjects. Subjects will be allocated to one of 2 dosing cohorts. Each cohort will have 12 subjects with 9 subjects randomised to receive AX-024.HCl and 3 subjects randomised to receive placebo.

There will be a data review following each dose level. Dose administration in the subsequent cohorts will only proceed after satisfactory data review on the blinded safety data and plasma PK data in the previous cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a body mass index (BMI) of 18 - 35 kg/m2, inclusive. BMI = Body weight (kg) / [Height (m)]2.
* Subjects must not be vegetarians or consume abnormal diets.
* Subject with no clinically significant abnormal serum biochemistry, haematology coagulation (Part B only) and urine examination values within 21 days of the first dose.
* Subject with a negative urinary drugs of abuse screen, determined within 21 days of the first dose (N.B. a positive alcohol result may be repeated at the discretion of the Investigator).
* Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 21 days of the first dose.
* Subject with no history of autoimmune disease, cardiac disease, kidney disease or any food intolerance.
* Male subject willing to use 2 effective methods of contraception i.e. established method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from Day 1 until 3 months afterwards.
* Subjects must be available to complete the study (including follow-up visit).
* Subjects must satisfy a medical examiner about their fitness to participate in the study
* Subjects must provide written informed consent to participate in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | 10 days
  Physical status (Vital signs; 12-lead ECG; Urinalysis; Haematology and biochemistry)

SECONDARY OUTCOMES:
maximal concentration (Cmax) | PK collected at multiple visits during the 10 days of treatment
Area under the plasma concentration versus time curve (AUC) | PK collected at multiple visits during the 10 days of treatment
Time to reach steady state | PK collected at multiple visits during the 10 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, Cardiff Road, United Kingdom